CLINICAL TRIAL: NCT02882919
Title: Improving Teen Health With Health Information Technology
Brief Title: Check Yourself v2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolyn McCarty (Other)
Responsible Party: Sponsor-Investigator, Carolyn McCarty, Research Associate Professor of Pediatrics, University of Washington and Investigator, Seattle Children's Research Institute, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01HS023383-01 (AHRQ)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Check Yourself v2.0 (Experimental): In the intervention group, adolescents complete Check Yourself which delivers personalized, motivational feedback on their health behaviors prior to their primary care appointment. Key components of Check Yourself include the provision of age normative feedback, goal setting strategies, and strategies to highlight discrepancies. Primary care providers will receive a summary report of health risk behaviors prior to their adolescent patient's primary care appointment.
  Interventions: Behavioral: Check Yourself v2.0
- Usual care (No Intervention): In the usual care group, patients are asked to complete health risk screening on a computer. No personalized feedback is provided to adolescents and primary care providers do not receive a summary report of the adolescent's health risk behaviors

INTERVENTIONS:
Behavioral: Check Yourself v2.0 — In the intervention group, adolescents complete Check Yourself which delivers personalized, motivational feedback on their health behaviors prior to their primary care appointment. Key components of Check Yourself include the provision of age normative feedback, goal setting strategies, and strategies to increase motivation for healthy behaviors. Primary care providers will receive a summary report of health risk behaviors prior to their adolescent patient's primary care appointment.
  Arms: Check Yourself v2.0

SUMMARY:
Health risk screening in adolescent primary care is infrequently performed and results are rarely followed by targeted intervention. In response to the need for screening-linked interventions, the study team has developed and optimized a web-based, electronic Personalized Motivational Feedback tool referred to as "Check Yourself v2.0" Based on motivational interviewing, a technique to mobilize personal change, Check Yourself is designed to promote healthy choices for the multiple behaviors relevant to adolescents.

DETAILED DESCRIPTION:
The proposed study is a randomized controlled trial that compares the effectiveness of Check Yourself v2.0 to usual care. The purpose of this study is to determine the impact of Check Yourself on reducing health risk behaviors and improving quality of care among adolescents receiving primary health care services relative to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Eligible adolescent participants will be13-18 years of age
* Able to understand English.
* Will have an appointment (or have a child with an appointment) with a participating medical practice.

Exclusion Criteria: Adolescents will be excluded from the study

* Participants do not meet age requirements
* Do not have an appointment with a participating provider at a PSPRN clinic,
* Lack the means to complete follow-up interviews (i.e., have neither telephone nor internet access)
* Have a sibling who has been/is being enrolled in the study or have previously participated in our previous trial comparing Check Yourself to usual care
* Not able to understand English.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2016-10; Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Number of Health risk behaviors | 3 months
  The risk behavior scale includes 22 values: 0 (min) to 21 (max). Higher scores indicate a worse outcome. Endorsement of any of the following counts as 1 (moderate risk) or 2 (high risk) on the scale depending on response and participant: ≥2 sugar-sweetened beverages consumed during typical day; ≤3 servings fruits/vegetables consumed during typical day; ≤3 days with 60+ minutes exercise during typical week; texting while driving in past 3 months; ≤7 hrs of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; tobacco use; days alcohol consumption in last 30 days (risk based on age) and/or number of drinks per drinking episode (risk based on age & sex); days marijuana consumption in last 30 days (risk based on age) and/or other drug use in past 3 months; not using birth control during last sexual intercourse and/or not "always" using a condom; & score of ≥10 on PHQ-9 depression.
Sweetened Beverage Consumption | 3 months
  Adolescent self-reported sweetened beverages consumed in a typical day in past 3 months. The sweetened beverages scale includes 4 values: 0 (min), 1, 2, or 3+ (max) sweetened beverages per day. Higher scores mean a worse outcome.
Physical Activity | 3 month
  Adolescent self-reported days with >60 minutes of physical activity in an average week in past 3 months. The physical activity scale includes 8 values: 0 (min) to 7 (max). Higher scores mean a better outcome.
Sleep | 3 month
  Adolescent self-reported hours of sleep on a typical night in past 3 months. . The sleep scale includes 13 values: 0 (min) to 12+ (max) hours of sleep per night. Higher scores mean a better outcome.
Alcohol Consumption (frequency) | 3 month
  Adolescent self-reported number of days of alcohol consumption and number of drinks during a typical drinking episode in the prior month
Marijuana and/or Other Drug Consumption | 3 month
  Adolescent self-reported number of days using marijuana in the past month and/or other drugs used in past 3 months. Two questions were used for this category. The marijuana frequency scale includes 31 values: 0 (min) to 30 (max) days in the past month. Higher scores mean a worse outcome. Adolescent self-reported use of other drugs in the past 3 months. The other drug score includes 2 values: 0=no (min) and 1=yes (max). Higher scores mean a worse outcome.
Depression | 3 month
  Adolescent self-reported depression as measured on the nine item Patient Health Questionnaire in past 2 weeks. The PHQ-9 depression scale includes 28 values: 0 (min) to 27 (max). Higher scores mean a worse outcome.
Seat belt Use | 3 month
  Adolescent self-reported frequency of seat belt use in a car in past 3 months. . The seatbelt use scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a better outcome.
Helmet Use | 3 month
  Adolescent self-reported frequency of helmet use while bicycling in past 3 months. The helmet use scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a better outcome.
Texting while driving | 3 month
  Adolescent self-reported endorsement of texting while driving in past 3 months. This question is only asked among adolescents who drive a car. The texting while driving scale includes 4 values: 1=never (min), 2=sometimes, 3=usually, or 4=always (max). Higher scores mean a worse outcome.
Condom Use and/or Birth Control Use | 3 month
  Adolescent self-reported condom use with sexual intercourse in past 3 months and/or use of birth control with last sexual intercourse. Two questions were used for this category. These questions were asked only to sexually active youth. The condom use scale includes 4 values: 1=always (min), 2=often, 3=sometimes, 4=never (max). Higher scores mean a worse outcome. The birth control scale includes 2 values: 0=no (min), 1=yes (max). Higher scores mean a better outcome.
Driving with Impairment | 3 month
  Adolescent self-reported driving under the influence of a substance in past 3 months. This question was asked only of adolescents who drive a car. The driving with impairment scale includes 2 values: 0=no (min) and 1=yes (max). Higher scores mean a worse outcome
Fruit and Vegetable Consumption | 3 month
  Adolescent self-reported fruits and vegetables consumed in a typical day in past 3 months. The fruits and vegetables scale includes 6 values: 0 (min), 1, 2, 3, 4, or 5+ (max). Higher scores mean a better outcome.
Percent of risk behaviors counseled on during primary care appointment | 1 day
  Percent of adolescent-reported health risk behaviors discussed with the healthcare provider during the primary care visit adjusted for the total number of health risk behaviors reported at baseline.
Adolescent Satisfaction with Care | 1 day
  Adolescent satisfaction with care will be assessed using 1 item adapted from the consumer Assessment Of healthcare Providers and Systems (CAHPS) measure at 1 day follow up. The CAHPS scale includes 10 values: 1 (min) to 10 (max). Higher scores mean a better outcome.
Tobacco Use | 3 month
  Adolescent self-reported endorsement of tobacco use in past 3 months. The tobacco use scale includes 2 values: 0=no (min) or 1=yes (max). Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Number of Health risk behaviors | 6 months
  Adolescent total count health-risk behaviors at 6 month follow-up including: During typical day: ≥2 sugar-sweetened beverages consumed and ≤3 servings fruits/vegetables consumed; ≤3 days with 60+ minutes exercise during typical week; having texted while driving in past 3 months; ≤7 hours of sleep during typical night; not "always" using seatbelt; not "always" using helmet when bicycling; having driven under the influence of substances; tobacco use; days of alcohol consumption in last 30 days (risk based on age: ≥1 day/30 days (ages 13-15), ≥2 days/30 days (ages 16-17), or ≥3 days/30 days (age 18)) and/or number of drinks per drinking episode (risk based on age and sex: ≥3 (Girls 13-17; Boys 13), ≥4 (Girls 18; Boys 14-15), or ≥5 (Boys 16-18)); days marijuana consumption in 30 day (risk based on age) and/or other drugs use in past 3 months; not using birth control during last sexual intercourse and/or not "always" using a condom; and score of ≥10 on PHQ-9.
Sweetened Beverage Consumption | 6 month
  Adolescent self-reported sweetened beverages consumed in a typical day in past 3 months
Fruit and Vegetable Consumption | 6 month
  Adolescent self-reported fruits and vegetables consumed in a typical day in past 3 months
Physical Activity | 6 month
  Adolescent self-reported days with >60 minutes of physical activity in an average week in past 3 months
Sleep | 6 month
  Adolescent self-reported hours of sleep on a typical night in past 3 months
Alcohol Consumption | 6 month
  Adolescent self-reported number of days of alcohol consumption and number of drinks during a typical drinking episode in the prior month
Marijuana and/or Other Drug Consumption | 6 month
  Adolescent self-reported number of days using marijuana in the past month and/or other drugs used in past 3 months
Depression | 6 month
  Adolescent self-reported depression as measured on the nine item Patient Health Questionnaire in past 2 weeks
Seat-belt Use | 6 month
  Adolescent self-reported frequency of seatbelt use in a car in past 3 months
Helmet Use | 6 month
  Adolescent self-reported frequency of helmet use while bicycling in past 3 months
Texting while driving | 6 month
  Adolescent self-reported endorsement of texting while driving in past 3 months
Condom Use and or Birth Control Use | 6 month
  Adolescent self-reported condom use with sexual intercourse in past 3 months and/or use of birth control at last sexual intercourse
Driving with Alcohol Impairment | 6 month
  Adolescent self-reported driving under the influence of a substance
Interval Receipt of Care | 3 months
  Dichotomous variable indicating receipt of any follow-up care to address risk behaviors identified at baseline adjusted for baseline number of health risk behaviors
Interval Receipt of Care | 6 months
  Dichotomous variable indicating receipt of any follow-up care to address risk behaviors identified at baseline adjusted for baseline number of health risk behaviors
Readiness to Change Ruler | 1-day
  Assessment of adolescent reported motivation to change overall health
Readiness to Change Ruler | 3 months
  Assessment of adolescent reported motivation to change overall health
Readiness to Change Ruler | 6 months
  Assessment of adolescent reported motivation to change overall health
Adolescent Health Self -Efficacy | 1 day
  Self-report of adolescent health self efficacy
Tobacco Use | 6 month
  Adolescent self-reported endorsement of tobacco use in past 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richardson L, Parker EO, Zhou C, Kientz J, Ozer E, McCarty C. Electronic Health Risk Behavior Screening With Integrated Feedback Among Adolescents in Primary Care: Randomized Controlled Trial. J Med Internet Res. 2021 Mar 12;23(3):e24135. doi: 10.2196/24135. PMID 33709942